CLINICAL TRIAL: NCT05654857
Title: The Prevalence of Family-unit Helicobacter Pylori Infection in Jiangsu Based on Non-invasive PCR in Stool
Brief Title: The Prevalence of Family-unit Helicobacter Pylori Infection in Jiangsu
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Zhenyu Zhang, Director of Gastroenterology, Nanjing First Hospital, Nanjing Medical University
Other Study IDs: KY20221124-09
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Helicobacter Pylori Infection
Keywords: Resistance Mutation; Fecal Drug Resistance Gene Detection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — stool specimen produced by normal excretion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PCR test in the stool — Patients will receive a prescription for a stool self-collection kit . Only the result of the PCR test in the stool will be considered for this arm. A positive test will determine Hp infection and the indication for treatment.

SUMMARY:
To assess Family-unit Helicobacter Pylori Infection rates and antimicrobial resistance rates in Jiangsu,China

DETAILED DESCRIPTION:
The study is a sample survey of the community population in cities of Jiangsu where the centers are located.The Helicobacter pylori infection and drug-resistant gene mutations are detected by real-time PCR performed on the stools of subjects.

ELIGIBILITY:
Inclusion Criteria:

1. community population
2. Fecal samples can be obtained, and the sample volume meets the requirements of the collection tube instructions
3. Only one person per family can be selected
4. Voluntarily participated in this study and signed an informed consent form

Exclusion Criteria:

1. The collector does not cooperate or has poor compliance;
2. Adequate and qualified fecal samples could not be obtained;
3. Stool samples were collected during diarrhea or constipation;
4. Antibiotics, bismuth preparations, proton pump inhibitors and other Hp sensitive drugs have been used within one month.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study was a sample survey of the community population in each central lock-in area, rather than hospital patients.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
The Prevalence of Family-unit Helicobacter Pylori Infection in Jiangsu | 2022.12.1-2023.6.30
  the Helicobacter Pylori Infection rate in Jiangsu family

SECONDARY OUTCOMES:
Trends of Antimicrobial Resistance of Helicobacter Pylori in Jiangsu | 2022.12.1-2023.6.30
  resistance to antimicrobial agents applicable for H. pylori eradication

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyu Zhang, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (16):
- China (16):
  - Changzhou Traditional Chinese medical hospital,Affiliated to Nanjing University of Chinese Medicine, Changzhou, Jiangsu
  - JinHu county people's hospital, Huaian, Jiangsu
  - The 1st people's hospital of Lianyungang, Lianyungang, Jiangsu
  - Nanjing First Hospital, Nanjing Medical University, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Rudong County People's Hospital, Nantong, Jiangsu
  - The Affiliated Shuyang Hospital of Xuzhou Medical University, Suqian, Jiangsu
  - Changshu No.1 People's Hospital, Suzhou, Jiangsu
  - Department of Gastroenterology Wuxi People's Hospital Affiliated to Nanjing Medical University, Wuxi, Jiangsu
  - The First People's Hospital of Xuzhou, Xuzhou Municipal Hospital Affiliated to Xuzhou Medical University, Xuzhou, Jiangsu
  - Dongtai People's Hospital, Yancheng, Jiangsu
  - Yancheng First Hospital Affiliated Hospital of Nanjing University Medical School, Yancheng, Jiangsu
  - Affiliated Hospital of Yangzhou University, Yangzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Changshu Hospital Affiliated to Nanjing University of Chinese Medicine, Suzhou
  - People's hospital of Yangzhong City, Zhenjiang

IPD SHARING:
Plan to Share IPD: No